CLINICAL TRIAL: NCT04189081
Title: A Clinical Study to Evaluate Dry Mouth Relief After Using an Experimental Mouth Rinse Compared to a Water Control
Brief Title: Improvement of Dry Mouth Sufferers After Using an Experimental Dry Mouth Rinse Compared to a Water Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSD2019158
Record Dates: First submitted 2019-12-04; First posted 2019-12-06 (Actual); Results first posted 2021-05-06 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Dry Mouth
MeSH Terms: conditions — Xerostomia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Experimental Mouth Rinse (Experimental): dry mouth rinse to be taken up to 5x a day, at least twice a day, 15 ml for 30 seconds for a week. Subjects will be restricted from using mouth rinse, acclimation products, eating or drinking for 6-hours after first use (at-home) on Day 1 and Day 8. There are no eating or drinking restrictions Day 2-Day 7.
  Interventions: Device: dry mouth rinse
- Water Control (Sham Comparator): Water will be used as a mouth rinse and can be taken up to 5x a day, at least twice a day, 15 ml for 30 seconds for a week. Subjects will be restricted from using water, acclimation products, eating or drinking for 6-hours after first use (at-home) on Day 1 and Day 8. There are no eating or drinking restrictions Day 2-Day 7.
  Interventions: Other: Water Control
- Positive Control (Active Comparator): dry mouth rinse to be taken up to 5x a day, at least twice a day, 15 ml for 30 seconds for a week. Subjects will be restricted from using mouth rinse, acclimation products, eating or drinking for 6-hours after first use (at-home) on Day 1 and Day 8. There are no eating or drinking restrictions Day 2-Day 7.
  Interventions: Device: dry mouth rinse

INTERVENTIONS:
Device: dry mouth rinse — relieves dry mouth symptoms by physically coating oral mucosal surfaces.
  Arms: Experimental Mouth Rinse; Positive Control
Other: Water Control — negative control
  Arms: Water Control

SUMMARY:
The objective of this study is to evaluate dry mouth relief in subjects with self-reported feeling of dry mouth after using an experimental mouth rinse or a positive control compared to a water control.

DETAILED DESCRIPTION:
This is a controlled, randomized, 3-treatment, parallel study for subjects with self-reported dry mouth symptoms as determined by an Oral Examination and subject responses to the Dry Mouth Inventory (DMI) questionnaire (see section 12) at the Acclimation visit. Qualified subjects will be randomly assigned to one of three treatments at the Baseline visit. Safety will be assessed by Oral Examinations at Baseline/Day1 and Day 8. Subjects will complete questionnaires before product use, immediately after product use (Day 1 only), and after 30 minutes, 1 hour, 2 hours, 4 hours and 6 hours of product use on Baseline/Day 1 and Day 8. The PPAQ II questionnaire will be completed on the morning of Day 8 (see study schedule for details).

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent prior to participation and be given a signed copy of the informed consent form;
* Sign a Confidentiality Disclosure Agree(CDA) form and be given a signed copy;
* Be at least 18 years of age;
* Agree not to participate in any other oral care studies for the duration of this study;
* Agree to delay elective dentistry, including dental prophylaxis, until study completion, and to report any non-study dentistry received during the course of the study;
* Agree to refrain from the use of any non-study oral hygiene products for the study duration including mouth rinse and toothpaste (flossing is permitted if part of their normal routine);
* Self-report a dry mouth feeling according to the modified DMI questions (Subject must answer at least 2 out of 4 questions with 'agree a little,' 'agree' or 'strongly agree');
* Agree to refrain from eating, drinking, smoking, using oral care products, using tobacco, using a medicated lozenge, chewing gum, or breath mints during the 6-hour test period (except snack after 4-hour Questionnaire);
* Agree to return for all scheduled visits and to follow all study procedures.

Exclusion Criteria:

* Any condition or disease, as determined by the Investigator/Designee, that could be expected to interfere with examination procedures, with compliance, or with the subject's safe completion of the study;
* Severe periodontal disease, as characterized by purulent exudate, generalized mobility, and/or severe recession;
* Active treatment for periodontitis;
* Having a history of allergies or hypersensitivity to mouth rinse or ingredients in commercial dental products or cosmetics;
* Self-reported pregnancy or the intent to become pregnant during the study, or breast feeding;
* Full or partial dentures or any orthodontic appliances such as braces or aligners, or tongue or mouth piercing;
* Inability to undergo any study procedure;
* Having untreated oral mucosal disease which in the opinion of the investigator could interfere with the study (e.g., current oral ulceration); or
* Evidence of gross intra-oral neglect or need for extensive dental therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2020-05-13 (Actual); Primary Completion 2020-07-08 (Actual); Study Completion 2020-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Milleman, DDS, Principal Investigator — Procter and Gamble
Locations (1):
- Salus Research, Fort Wayne, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Self-reported a dry mouth feeling according to the modified DMI questions (Subject must have answered at least 2 out of 4 questions below with 'agree a little,' 'agree' or 'strongly agree'):
  How much do you agree or disagree that you experience the following? (strongly disagree, disagree, disagree a little, agree a little, agree, strongly agree)
  1. No moisture in the mouth
  2. Lips sticking to teeth
  3. Tongue sticking to roof of mouth
  4. Throat feels dry
Period: Overall Study
Arm/Group | Water Control | Experimental Mouth Rinse | Positive Control
Started | 46 | 45 | 46
Completed | 45 | 45 | 45
Not Completed | 1 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Water Control | Experimental Mouth Rinse | Positive Control | Total
Number analyzed (Participants) | 46 | 45 | 46 | 137
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (11.83) | 56.2 (14.97) | 58.3 (12.04) | 57.6 (12.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 37 | 37 | 113
  Male | 7 | 8 | 9 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 2
  Not Hispanic or Latino | 45 | 44 | 46 | 135
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 7 | 12 | 22
  White | 41 | 38 | 33 | 112
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Response to "Relieving the Discomfort of Dry Mouth" From the Modified PPAQ I 4- and 6-hours Post-use on Day 1 of Treatment
Description: Product Performance and Attributes (PPAQ I)
  Since you have been using the product, please rate each of the following at this timepoint: (Select one response for attribute)- excellent=5, very good=4, good=3, fair=2, poor=1:
  1) Relieves the discomfort of your dry mouth
Time Frame: 4-hours
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Water Control | Experimental Mouth Rinse | Positive Control
Number analyzed (Participants) | 46 | 45 | 46
score on a scale | 2.51 (0.158) | 3.26 (0.160) | 3.43 (0.158)

2. Primary Outcome: Response to "Relieving the Discomfort of Dry Mouth" From the Modified PPAQ I 4- and 6-hours Post-use on Day 1 of Treatment
Description: as for outcome 1
Time Frame: 6-hours
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Water Control | Experimental Mouth Rinse | Positive Control
Number analyzed (Participants) | 46 | 45 | 46
score on a scale | 2.70 (0.154) | 3.46 (0.156) | 3.36 (0.154)

ADVERSE EVENTS:
Time Frame: Products were used over 8 days
Description: investigator/examiner observed
Arm/Group | Water Control | Experimental Mouth Rinse | Positive Control
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/45 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/45 | 0/46
Other Adverse Events (participants affected / at risk) | 3/46 | 2/45 | 2/46
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Water Control (N=46) | Experimental Mouth Rinse (N=45) | Positive Control (N=46)
mouth injury (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 1 (1)
Aphthous Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI agreed to not publish results without prior written consent of Sponsor.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-01): https://cdn.clinicaltrials.gov/large-docs/81/NCT04189081/Prot_SAP_000.pdf